CLINICAL TRIAL: NCT07041801
Title: Phase I/II Clinical Study on the Safety, Efficacy, Pharmacodynamics and Immunogenicity of Human Umbilical Cord Mesenchymal Stem Cell Injection (hUCMSCs) in the Treatment of Patients With Moderate to Severe Systemic Lupus Erythematosus
Brief Title: Treatment of Systemic Lupus Erythematosus With Human Umbilical Cord Mesenchymal Stem Cells
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK-SLE-I/01
Record Dates: First submitted 2025-04-27; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- hUC-MSCs treatment (low dose) (Experimental): Conventional plus hUC-MSCs treatment (low dose)
  Interventions: Drug: hUC-MSCs treatment (low dose)
- hUC-MSCs treatment （medium dose） (Experimental): conventional therapy plus hUC-MSCs treatment （medium dose）
  Interventions: Biological: hUC-MSCs treatment (medium dose)
- hUC-MSCs treatment （high dose） (Experimental): conventional therapy plus hUC-MSCs treatment （high dose）
  Interventions: Biological: hUC-MSCs treatment (high dose)
- hUC-MSCs treatment （Double dose） (Experimental): conventional therapy plus hUC-MSCs treatment（Double dose）
  Interventions: Biological: hUC-MSCs treatment （Double dose）
- Placebo (Placebo Comparator): conventional therapy plus Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hUC-MSCs treatment (low dose) — patients will receive conventional therapy plus low dose hUC-MSCs treatment,The dosage is 1E6 cells/kg.
  Arms: hUC-MSCs treatment (low dose)
Biological: hUC-MSCs treatment (medium dose) — patients will receive conventional therapy plus medium dose hUC-MSCs treatment,The dosage is 3E6 cells/kg.
  Other Names: MSC-medium
  Arms: hUC-MSCs treatment （medium dose）
Biological: hUC-MSCs treatment (high dose) — patients will receive conventional therapy plus high dose hUC-MSCs treatment,The dosage is 5E6 cells/kg.
  Other Names: MSC-high
  Arms: hUC-MSCs treatment （high dose）
Drug: Placebo — patients will receive conventional therapy plus Placebo
  Arms: Placebo
Biological: hUC-MSCs treatment （Double dose） — Double dosing is selected by the investigators and the sponsor based on the data from the single-dose part of the study. One superior dose is chosen for multiple dosing (tentatively set at 3E6 cells/kg, administered twice with an interval of 4 weeks; the actual dose, frequency and interval of multiple dosing can be adjusted according to the available data). During the trial, stable standard treatment is allowed.
  Arms: hUC-MSCs treatment （Double dose）

SUMMARY:
This study will investigate the safety and efficacy of allogeneic umbilical cord-derived stem cell therapy in treating patients with moderate to severe systemic lupus erythematosus.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Fully understand the purpose, nature, methods of the trial, as well as possible adverse reactions, voluntarily participate as a subject, and sign the informed consent form.
2. Age 18-65 years old (inclusive of the boundaries, based on the date of signing the informed consent form), regardless of gender;
3. The subjects (both male and female) must agree not to have a reproductive plan during the trial period and after the injection administration for at least 12 months, and voluntarily take effective contraceptive measures with their partners (see Appendix 1), and have no plans for sperm donation or egg donation;
4. According to the diagnostic classification criteria of the European League Against Rheumatism (EULAR) and the American College of Rheumatology (ACR) in 2019, diagnosed with systemic lupus erythematosus (SLE);

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, nature, methods of the trial and possible adverse reactions, voluntarily become a subject, and sign the informed consent form.
2. Age 18-65 years old (inclusive of the boundary values, based on the time of signing the informed consent form), no gender restrictions;
3. The subjects (male and female) must agree not to have a reproductive plan during the trial period and after the injection administration for at least 12 months, and voluntarily take effective contraceptive measures with their partners (see Appendix 1), and have no plans for sperm donation or egg donation;
4. According to the diagnostic classification criteria of the European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) in 2019, diagnosed with systemic lupus erythematosus (SLE);
5. Meet one of the following conditions: the antinuclear antibody (ANA) is positive at 1:80 during screening or the anti-dsDNA antibody is positive during screening or the anti-Sm antibody is positive during screening;

Exclusion Criteria:

1. Those who are judged by the researchers to be likely to be allergic to the investigational drug or any component thereof;
2. Those who have had central nervous system diseases within 8 weeks before administration (including but not limited to epilepsy, mental illness, interstitial encephalopathy syndrome, stroke, encephalitis, central nervous system vasculitis, etc.);
3. Those who have undergone major organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplantation;
4. Those who have any major diseases/diseases or unstable clinical conditions (such as liver, kidney, hematological, endocrine, pulmonary, immune, mental, etc.) or active infections/infectious diseases with evidence, and according to the researchers' clinical judgment, if the subjects participate in the study, it will significantly increase the risks for the subjects;
5. Those who currently have known or suspected malignant tumors;
6. Those who have severe pulmonary arterial hypertension (>70 mmHg, 1 mmHg = 0.133 kPa), or mild to moderate pulmonary arterial hypertension patients with severe cardiopulmonary insufficiency;
7. Those who have antiphospholipid syndrome (APS), or have a history of catastrophic antiphospholipid syndrome (CAPS), or although not diagnosed as APS, but are evaluated by the researchers as having an increased risk of thrombosis;
8. Those who have herpes zoster infection within 90 days before administration, or any infection that requires hospitalization treatment or intravenous or intramuscular injection of antibiotics within 60 days before administration;
9. Those who have undergone major surgical operations within 28 days before administration, or those who are expected to undergo major surgical operations during the trial;
10. Subjects who have positive serological tests for viral hepatitis during the screening period, positive human immunodeficiency virus antibody (HIV-Ab), positive hepatitis B surface antigen (HBsAg), positive hepatitis C antibody (HCV-Ab), or positive Treponema pallidum antibody (TP-Ab);
11. Other situations that the researchers consider may affect the subjects' willingness to provide informed consent or follow the trial protocol, or situations where the subjects' participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2027-09-05 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | day 1 to day 28
  Analysis for the primary endpoint will be descriptive in nature. safety and tolerability will be measured by the number of AEs and SAEs observed. Adverse event incidents will be summarized descriptively. The severity grade of each recorded AE, and their relationship to study treatment will be analyzed. The action taken and outcome will also be analyzed accordingly.

SECONDARY OUTCOMES:
Efficacy Endpoint | The 24th week after administration of the test drug.
  The proportion of subjects whose SLEDAI-2000 score (a scale for assessing the disease activity of systemic lupus erythematosus) decreased by ≥ 4 points Total score ranging from 0 to 105.
  Interpretation: Scores are categorized to indicate disease activity:
  0: No activity 1-5: Mild activity 6-10: Moderate activity 11-19: High activity
  ≥20: Very high activity
  Improvement is defined as a decrease in score.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Beike Bio-Technology Co. Ltd., Shenzhen, Guangdong, China